CLINICAL TRIAL: NCT06694753
Title: A Phase 1, Placebo-controlled, Blinded, Dose-escalation Study to Evaluate the Safety and Immunogenicity of mRNAs Encoding HIV Immunogens (eOD-GT8 60mer, Core-g28v2 60mer, N332-GT5 gp151) in Adult Participants Without HIV and in Overall Good Health in South Africa.
Brief Title: Safety and Immunogenicity Study of Three mRNAs Encoding HIV Immunogens in Adult Participants Without HIV and in Overall Good Health in South Africa.
Acronym: IAVI G004
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: ModernaTX, Inc. (Industry); The Scripps Research Institute (Other); National Institute of Allergy and Infectious Diseases (NIAID)/Division of AIDS (DAIDS) (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DESIIGN001/ IAVI G004
Record Dates: First submitted 2024-11-05; First posted 2024-11-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Cohorts 1A and 2A in Part A will be enrolled concurrently. Randomization to study product or placebo will take place within each cohort. After Part A is fully enrolled, there will be a planned safety hold to review all safety data from participants for one month following the final participant's first vaccination (week 0) in Part A. Enrollment in Part B will not proceed without the formal approval of the Protocol Safety Review Team (PSRT). Similar to enrollment in Part A, Cohorts 1B and 2B in Part B will be enrolled concurrently. Randomization to study product or placebo will take place within each cohort.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study team will be blinded to treatment assignment within a cohort but not across cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Cohort 1A Group 1: mRNA-1645-eODGT8 + mRNA-1645-CoreG28v2 (Experimental): Participants will receive one injection of 10 mcg mRNA-1645-eODGT8 to be administered as a 0.5 mL IM injection into the deltoid at Week 0 and one injection of 10 mcg mRNA-1645-CoreG28v2 to be administered as a 0.5 mL IM injection into the deltoid at Week 8.
  Interventions: Biological: mRNA-1645-eODGT8; Biological: mRNA-1645-CoreG28v2
- Cohort 1A Group 2: Placebo (Placebo Comparator): Participants will receive 0.9% sodium chloride to be administered as a 0.5-mL IM injection into the deltoid at Weeks 0 and 8.
  Interventions: Biological: Placebo
- Cohort 2A Group 3: mRNA-1645-N332GT5 (Experimental): Participants will receive 10 mcg of mRNA-1645-N332GT5 to be administered as a 0.5 mL IM injection into the deltoid at Weeks 0 and 8.
  Interventions: Biological: mRNA-1645-N332GT5
- Cohort 2A Group 4: Placebo (Placebo Comparator): Participants will receive 0.9% sodium chloride to be administered as a 0.5-mL IM injection into the deltoid at Week 0 and Week 8.
  Interventions: Biological: Placebo
- Cohort 1B Group 5: mRNA-1645-eODGT8 + mRNA-1645-CoreG28v2 (Experimental): Participants will receive one injection of 30 mcg mRNA-1645-eODGT8 to be administered as a 0.5 mL IM injection into the deltoid at Week 0 and one injection of 30 mcg mRNA-1645-CoreG28v2 to be administered as a 0.5 mL IM injection into the deltoid at Week 8.
  Interventions: Biological: mRNA-1645-eODGT8; Biological: mRNA-1645-CoreG28v2
- Cohort 1B Group 6: Placebo (Placebo Comparator): Participants will receive 0.9% sodium chloride to be administered as a 0.5-mL IM injection into the deltoid at Week 0 and Week 8.
  Interventions: Biological: Placebo
- Cohort 2B Group 7: mRNA-1645-N332GT5 (Experimental): Participants will receive 30 mcg of mRNA-1645-N332GT5 to be administered as a 0.5 mL IM injection into the deltoid at Weeks 0 and 8.
  Interventions: Biological: mRNA-1645-N332GT5
- Cohort 2B Group 8: Placebo (Placebo Comparator): Participants will receive 0.9% sodium chloride to be administered as a 0.5-mL IM injection into the deltoid at Week 0 and Week 8.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1645-eODGT8 — eOD-GT8 60mer is a self-assembling nanoparticle composed of 60 subunits of the engineered HIV-1 gp120 outer domain germline targeting version 8 (eOD-GT8) fused to an engineered form of a bacterial enzyme, Lumazine Synthase, through a 15-amino acid Glycine-Serine linker. eOD-GT8 60mer will be delivered using an mRNA lipid nanoparticle (LNP) platform. To be administered by intramuscular (IM) injection at doses of 10 or 30 mcg.
  Other Names: eOD-GT8 60mer mRNA
  Arms: Cohort 1A Group 1: mRNA-1645-eODGT8 + mRNA-1645-CoreG28v2; Cohort 1B Group 5: mRNA-1645-eODGT8 + mRNA-1645-CoreG28v2
Biological: mRNA-1645-CoreG28v2 — core-g28v2 60mer is a nanoparticle composed of 60 protein subunits of an engineered core-gp120 fused to an engineered form of a bacterial enzyme, Lumazine Synthase, through a 21-amino acid Glycine-Serine linker. Core-g28v2 60mer will be delivered using an mRNA-LNP platform. To be administered by IM injection at doses of 10 or 30 mcg.
  Other Names: core-g28v2 60mer mRNA
  Arms: Cohort 1A Group 1: mRNA-1645-eODGT8 + mRNA-1645-CoreG28v2; Cohort 1B Group 5: mRNA-1645-eODGT8 + mRNA-1645-CoreG28v2
Biological: mRNA-1645-N332GT5 — N332-GT5 gp151 is an HIV envelope glycoprotein gp151 trimer based on BG505 SOSIP MD39 (clade A) trimer with "germline-targeting" mutations added that confer the ability to bind germline precursors of BG18 class B cells. N332-GT5 gp151 will be delivered using an mRNA-LNP platform. To be administered by IM injection at doses of 10 or 30 mcg.
  Other Names: N332-GT5 gp151 mRNA
  Arms: Cohort 2A Group 3: mRNA-1645-N332GT5; Cohort 2B Group 7: mRNA-1645-N332GT5
Biological: Placebo — Saline
  Other Names: Saline; Diluent
  Arms: Cohort 1A Group 2: Placebo; Cohort 1B Group 6: Placebo; Cohort 2A Group 4: Placebo; Cohort 2B Group 8: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of mRNAs encoding HIV immunogens (eOD-GT8 60mer, core-g28v2 60mer, N332-GT5 gp151) in adult participants without HIV and in overall good health in South Africa.

DETAILED DESCRIPTION:
This study will evaluate the safety and immunogenicity of 3 experimental HIV vaccines in adult participants without HIV and in overall good health in South Africa. The study vaccines are called mRNA-1645-eODGT8, mRNA-1645-CoreG28v2 and mRNA-1645-N332GT5.

The study will be conducted in two parts (Part A and B). Part A will include two Cohorts, each with 2 groups: Cohort 1A Group 1, Cohort 1A Group 2, Cohort 2A Group 3, and Cohort 2A Group 4. Part B will include two Cohorts, each with 2 groups: Cohort 1B Group 5, Cohort 1B Group 6, Cohort 2B Group 7, and Cohort 2B Group 8.

Participants in Part A Cohort 1A will be randomly assigned to receive mRNA-1645-eODGT8 followed by mRNA-1645-CoreG28v2 or to receive placebo. Participants in Part A Cohort 2A will be randomly assigned to receive two doses of the mRNA-1645-N332GT5 vaccine or to receive placebo. Cohorts 1A and 2A in Part A will be enrolled concurrently, and randomization to study product or placebo will take place in each cohort. Depending on their group, participants will receive 10 mcg of mRNA-1645-eODGT8, mRNA-1645-N332GT5 or Placebo by injection at Week 0 and 10 mcg of mRNA-1645-CoreG28v2, mRNA-1645-N332GT5, or Placebo at Week 8.

Participants in Part B Cohort 1B will be randomly assigned to receive an increased dose of the mRNA-1645-eODGT8 and mRNA-1645-CoreG28v2 vaccine or to receive placebo. Participants in Part B Cohort 2B will be randomly assigned to receive an increased dose of the mRNA-1645-N332GT5 vaccine or to receive placebo. Cohorts 1B and 2B in Part B will be enrolled concurrently, and randomization to study product or placebo will take place in each cohort. Depending on their group, participants will receive 30 mcg of mRNA-1645-eODGT8, mRNA-1645-N332GT5 or Placebo by injection at Week 0 and 30 mcg of mRNA-1645-CoreG28v2, mRNA-1645-N332GT5, or Placebo at Week 8.

Additional study visits will occur at Weeks 2, 7.5, 10, 15.5, and 24. Study visits may include physical examinations, medical history, vaccine injections, blood and urine collection, electrocardiogram, leukapheresis, lymph node cell collection, pregnancy test, HIV testing, risk reduction counseling, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrates an understanding of the study and is able and willing to complete the informed consent process.
2. 18 to ≤ 55 years old, on day of enrollment.
3. Available for clinic follow-up through the last clinic visit.
4. Willingness to undergo FNA and leukapheresis.
5. Agrees not to enroll in another study of an investigational agent during participation in the trial. If a potential participant is already enrolled in another clinical trial, approvals from the other trial Sponsor and the IAVI Medical Monitor are required prior to enrollment into DESIIGN001/IAVI G004.
6. In good general health according to the clinical judgment of the Investigator.
7. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgment of the Investigator.
8. Assessed by clinical staff as having a low likelihood of acquiring HIV per guidelines (see Appendix 4), agrees to discuss their potential for HIV acquisition, agrees to prevention counseling, and agrees to avoid behaviors associated with a higher likelihood of acquiring HIV through the final study visit. "Low likelihood" may include persons stably taking pre-exposure prophylaxis (PrEP) as prescribed in Appendix 4.
9. Hemoglobin (Hgb):

   * ≥12.0 g/dL for AFAB volunteers
   * ≥13.0 g/dL for cisgender AMAB volunteers or for volunteers who have been on masculinizing hormone therapy for more than 6 consecutive months
   * ≥12.0 g/dL for AMAB volunteers who have been on feminizing hormone therapy for more than 6 consecutive months
   * For volunteers who have been on gender-affirming hormone therapy for less than 6 consecutive months, determine Hgb eligibility based on their sex assigned at birth.
10. White blood cell (WBC) count = 2,500 to 12,000/mm3.
11. Platelets = 125,000 to 550,000/mm3.
12. Alanine aminotransferase (ALT) <2.5 × upper limit of institutional reference range.
13. Serum creatinine ≤1.1× upper limit of normal (ULN) based on the institutional normal range.
14. Systolic blood pressure of 90 to <140 mmHg and diastolic blood pressure of 50 to <90 mmHg at the screening visit. The average blood pressure between the screening visit and the enrollment visit must be below 140 mmHg systolic and 90 mmHg diastolic. A single measurement ≥160 mmHg systolic or 100 mmHg diastolic during the current study evaluation is exclusionary.
15. Negative HIV test results by one of the following options:

    * A negative European Conformity (CE)-marked enzyme immunoassay (EIA)
    * A chemiluminescent microparticle immunoassay (CMIA)
    * A negative result on 2 HIV rapid tests (one of these rapid tests must be CE-marked)
16. Negative for anti-Hepatitis C virus (HCV) Abs (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV Abs are detected.
17. Negative for Hepatitis B surface antigen (HBsAg).
18. For volunteers AFAB or assigned intersex at birth who are capable of becoming pregnant (hereafter referred to as "persons of pregnancy potential"):

    * Must agree to use effective means of contraception from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination time point (see Appendix 5).
    * Must have a negative beta human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on day of enrollment.

    Note: Persons who are NOT of pregnancy potential due to total hysterectomy or bilateral oophorectomy or menopause (no menses for ≥1 year) are not required to undergo pregnancy testing.
19. Volunteers AFAB or assigned intersex at birth must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination time point.

Exclusion Criteria:

1. Volunteer is nursing or pregnant.
2. Body mass index (BMI) ≥40 kg/m2. Enrollment of individuals with BMI ≥40 kg/m2, whom the site investigator assesses are in good health, may be considered by the IAVI Medical Monitor.
3. Diabetes mellitus (DM). Type 2 DM controlled with diet alone (and confirmed by HgbA1c ≤7% within the last 6 months) or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with Type 2 DM that is well controlled on hypoglycemic agent(s) may be considered by the IAVI Medical Monitor on a case-by-case basis, provided that the HgbA1c is ≤8% within the last 6 months (CRC staff may draw these at screening).
4. Previous or current recipient of an investigational HIV vaccine (previous placebo/control recipients are not excluded).
5. Receipt of non-HIV investigational vaccine(s) received within the last 1 year. Exceptions include vaccines that have subsequently undergone licensure or Emergency Use Authorization (EUA) by the FDA or World Health Organization (WHO) Emergency Use Listing (EUL), or if outside the US, by the national Regulatory Authority authorizing this clinical trial.
6. Congenital or acquired immunodeficiency, including systemic medication use likely to impair immune response to vaccine in the opinion of the Investigator, such as glucocorticoid use, prednisone ≥10 mg/day within 3 months prior to enrollment.
7. Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires approval by the IAVI Medical Monitor.
8. Previous receipt of VRC01 or VRC07-523LS monoclonal antibody (mAb).
9. Receipt of any vaccine within 4 weeks prior to enrollment or planned receipt within 4 weeks of investigational vaccine administration.
10. History of myocarditis and/or pericarditis.
11. A past history of immune-mediated disease, including but not limited to thyroid disease, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, celiac disease, seronegative inflammatory arthritis, systemic sclerosis, and Type 1 diabetes (for other examples, see Appendix 8).
12. History of or active severe skin conditions, including, but not limited to, cutaneous mastocytosis, psoriasis, atopic dermatitis, lichen planus, hidradenitis suppurativa, bullous pemphigoid, and urticarial vasculitis.
13. Systemic or local conditions with urticaria as a manifestation, including urticarial vasculitis, maculo-papular cutaneous mastocytosis (formerly urticaria pigmentosa), mast cell activation syndrome, Gleich's syndrome (episodic angioedema with eosinophilia), Well's syndrome (granulomatous dermatitis with eosinophilia/eosinophilic cellulitis), bullous pemphigoid, or adult-onset Still's disease.
14. Receipt of antigen-based immunotherapy.
15. Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life of more than 7 days (or unknown half-life) within the past year, approval by the IAVI Medical Monitor is required for enrollment.
16. History of serious reaction (eg, hypersensitivity, anaphylaxis) to any vaccine or component of the study-vaccine regimen.
17. History of hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
18. History of urticaria and/or dermatographism.
19. History of atopy (diagnosed or confirmed by a clinician).
20. Bleeding disorder diagnosed by a clinician that would make study procedures a contraindication.
21. History of seizure(s) within the past 3 years, or if volunteer has used medications to prevent or treat seizure(s) at any time within the past 3 years.
22. Asplenia or functional asplenia.
23. Any other chronic or clinically significant condition that, in the clinical judgment of the Investigator, would jeopardize the safety or rights of the study participant, including but not limited to: clinically significant forms of substance use or alcohol use disorder(s), serious psychiatric disorders, any suicide attempt within the past 1 year (if between 1 and 2 years, consult the IAVI Medical Monitor for approval), or cancer that, in the clinical judgment of the Investigator, has potential for recurrence (excluding basal cell carcinoma).
24. Asthma (diagnosed or confirmed by a clinician).
25. History of allergy to local anesthetic (Novocaine, Lidocaine).
26. Investigator concern for difficulty with venous access based on clinical history and physical examination. For example, persons with a history of intravenous drug use or substantial difficulty with previous blood draws.
27. Has donated ≥450 mL of blood products within 28 days prior to the Screening Visit or plans to donate blood products within 28 days post study injection.
28. Is working or has worked as study personnel or is an immediate family member or house member of study personnel, study site staff, or Sponsor personnel.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-12-08 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess the incidence of local and systemic reactogenecity and treatment-emergent adverse events [Safety and Tolerability]. | Measured a minimum of 7 days following receipt of any study vaccination
  * Local and systemic reactogenicity signs and symptoms will be collected for a minimum of 7 days following receipt of any study vaccination.
  * AEs leading to early participant withdrawal or permanent discontinuation, SAEs, medically attended adverse events (MAAEs), and AESIs will be collected throughout the study. Additionally, all AEs will be collected for 30 days after any receipt of study vaccination.
To evaluate the induction of VRC01- or BG18-class IgG B cell responses by the vaccine regimens. | V01 [W0, baseline] V04 [W7.5, 7.5 wks. post 1st vacc.] V06 [W10, 2 wks. post 2nd vacc.] V07 [W15.5, 7.5 wks. post 2nd vacc.]
  • Proportion of vaccinees with VRC01- or BG18-class IgG B cells, and frequency of VRC01- or BG18-class B cells among IgG+ B cells in PBMCs or in germinal centers, at baseline and after each study product administration, as determined by B-cell phenotyping and BCR sequencing.

SECONDARY OUTCOMES:
To evaluate vaccine-specific and epitope-specific binding Ab responses elicited by the vaccine regimens. | Measured at baseline (at Week 0), 2 weeks post 1st vaccination (at Week 2), 7.5 weeks post 1st vaccination (at Week 7.5), 2 weeks post 2nd vaccination (at Week 10), and 7.5 weeks post 2nd vaccination (at Week 15.5)
  Response rate and magnitude of serum IgG binding Abs as assessed by BAMA at baseline and after each study product administration.

CONTACTS AND LOCATIONS:
Overall Officials: Linda-Gail Bekker, Principal Investigator — Desmond Tutu Health Foundation/Center, University of Cape Town
Locations (6):
- South Africa (6):
  - Setshaba Research Centre CRS, Soshanguve, Gauteng
  - Perinatal HIV Research Unit (PHRU), Soweto, Gauteng
  - CAPRISA eThekwini CRS, Durban, KwaZulu-Natal
  - Isipingo CRS, Isipingo, KwaZulu-Natal
  - Desmond Tutu Health Foundation Emavundleni CRS, Cape Town, Western Cape
  - Desmond Tutu Health Foundation- Groote Schuur Hospital/J52, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
A primary manuscript will be prepared after the data analysis is available and the results of the study will be published in searchable, peer reviewed scientific literature according to the, allowing unrestricted access and reuse of all peer-reviewed published research.Underlying, anonymized datasets will be made publicly available. The final clinical study report will be made available to the principal investigators. The Sponsor will also provide investigators with the full summary of the study results, which the investigators may share with the study participants and stakeholders, as appropriate.
Supporting Information: Study Protocol
Time Frame: No later than 12 months after the trial completion.
Access Criteria: The study data and documents will be shared publicly after the conclusion of the study and at the time of primary manuscript publication. Documentation will include; Study protocols, annotated CRFs and Statistical Analysis Plans. The datasets will be posted as SAS transport files XPT and as CSV files. IAVI will post packages to the Vivli online repository, accessible to the public by website. Vivli uses an independent peer review process to evaluate the validity of external requests.To protect participant privacy and comply with data protection laws, IAVI will utilize an independent organization who specializes in clinical trial data anonymization and privacy to prepare anonymized data packages for public consumption. Manuscripts will be made available at the time of publication through placement in apublicly available repository and openly licensed. Post-publication Data Packages wil be made available at publication in compliance with specific journal requirements.